CLINICAL TRIAL: NCT01187147
Title: Effects of Green Tea Extract (GTE) on Systemic Oxidative and Antioxidative Status in Chinese Patients With Stable Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: David CL Lam, University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HKCTR415
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-08

CONDITIONS: Asthma
Keywords: Asthma, green tea, antioxidants
MeSH Terms: conditions — Asthma | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Green Tea (Experimental): Recruited subjects will be asked to take green tea capsules for 3 months and then stopped for another 3 months.
  Interventions: Dietary Supplement: green tea extract

INTERVENTIONS:
Dietary Supplement: green tea extract — Green tea extract capsule, equivalent to 450 ml 2% Green tea containing 540mg EGCG/day
  Other Names: Lung Chen green tea

SUMMARY:
Asthma is a disease characterized by chronic inflammation in the airways. Recent research has demonstrated that one of the reasons for the chronic inflammatory state is an imbalance between oxidative stress and antioxidative defenses in patients with asthma.

Green tea is a common beverage consumed by Chinese patients from all walks of life. Green tea contains chemical components that are thought to have immunomodulatory actions in chronic inflammation.

The investigators propose to recruit 35 patients with stable asthma. Recruited subject will be given oral tablets containing Green tea extract (GTE) to be taken daily for three months. Clinical follow up and assessment will be done at baseline, on completion of GTE intake at three months, and at three months after GTE intake has been stopped. A questionnaire on their health status and the frequency of symptoms and use of bronchodilators and inhaled steroids will be completed, spirometry will be done and a venous blood sample will be taken during recruitment and during each reassessment at 3 and 6 months. Measurement of oxidants/antioxidants (GSH, GSSG, SOD, CAT and GPx) will be carried out on the blood samples. Oxidants/antioxidants will be compared and correlated with lung function results.

This study would provide us with pilot data as to whether GTE, a strong antioxidant with immunomodulatory actions, has any effect on reducing the oxidative stress and improving the antioxidant status in patients with asthma and whether these changes are accompanied improvement in clinical status.

Hypothesis Green tea extract (GTE) reduces oxidative stress and improves antioxidant defenses in Chinese patients with asthma

DETAILED DESCRIPTION:
1. Background

   Asthma constitutes a significant health problem both in Hong Kong and worldwide (1). Different risk factors for asthma have been identified. These include atopy (2), family history of asthma, exposure to indoor aeroallergens (3) air pollution (4) and exposure to environmental tobacco smoke (5).

   Asthma is associated with a chronic inflammatory state in the airway. The inflammatory component is thought to result from an imbalance between an increased free radical formation (oxidative stress) and a reduction of antioxidative defenses. Reactive oxygen species (ROS) such as superoxide radicals and hydrogen peroxide were found to be increased in patients with asthma indicating the presence of oxidative stress, and the increased level of ROS has also been found to correlate with asthma severity (6).

   The airway displays a wide range of enzymatic and non-enzymatic antioxidant defenses, including reduced glutathione (GSH), superoxide dismutase (SOD), catalase and glutathione peroxidase (GPx). There is evidence of reduced antioxidant defenses, namely GPx and SOD activity, in asthma patients (6). Furthermore, the measurement of the oxidized form of glutathione, (glutathione disulfide, GSSG) could be used as an index to reflect the degree of oxidative stress in asthma and the level of GSSG has been reported to be high in the bronchial washings of asthma patients (7). We have reported that patients with asthma showed significantly increased erythrocyte GSSG, SOD and catalase activities with concomitant reduction of erythrocyte GPx (8). These results indicate a state of increased oxidative stress accompanied by an altered state of systemic antioxidant status in asthma patients.

   Green tea represents one of the common beverages consumed by people from all walks of life. Epigallocatechin gallate (EGCG) is the major polyphenol (catechin) in green tea. Green tea extract (GTE) demonstrates anti-inflammatory and immunomodulatory activities. GTE has been shown to damp down neutrophil chemotaxis and attenuates interleukin-mediated inflammatory reaction cascades (9). It has also been shown to attenuate lung injury in experimental mouse model (10).

   This proposal is to investigate the effects of GTE on systemic oxidative and antioxidative status, and whether these changes are associated with changes in clinical status in local Chinese patients with stable asthma.
2. Research plan and methodology

Aims of the study

1. To determine and compare erythrocyte levels of GSSG, SOD, CAT and GPx in patients with asthma after 3 months of treatment with GTE and after GTE has been stopped for an equivalent period.
2. To determine and compare plasma levels of inflammatory marker C-reactive protein (CRP) and inflammatory mediators, interleukin-6 (IL-6) and IL-8 in these patients.

Study design This is an intervention study with patients serving as their own control

Material and Methods Patients

The investigators propose to recruit out-patients with asthma in stable clinical condition and have no acute asthmatic attack in the recent 3 months prior to recruitment. After initial assessment, recruited patients will be given GTE to be taken three times a day for 3 months. They will be reassessed at 3 months when GTE will be stopped and again at the end of 6 months. The clinical status and biochemical parameters when they are on GTE will be compared with similar parameters when they are not on GTE.

ELIGIBILITY:
Inclusion Criteria:

* Asthma patients being followed up in out-patient clinic with stable clinical condition.
* Age 18 - 70 years

Exclusion Criteria:

* Patients with known significant concomitant illness including pulmonary causes (COPD, pulmonary tuberculosis, lung cancer, bronchiectasis, interstitial lung disease and obstructive sleep apnoea) and non-pulmonary causes (hypertension, diabetes mellitus, ischaemic heart disease, stroke, cancer of other organ sites).
* Patients with unstable asthma
* Patients with alcohol dependence
* Patients with abnormal liver function or is a hepatitis B or C carrier,
* Patients who have habits of taking tea or tea extract, or under other clinical drug trial or herbs
* Patients who are pregnant or breast feeding
* Patients who are unwilling to participate or unable to give written consent on his/her own

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Serum Inflammatory markers | Six months
  Serum catalase, superoxide dismutase, glutathione peroxidase, oxidized glutathione and other inflammatory markers including CRP, IL6 and IL8

SECONDARY OUTCOMES:
Respiratory symptoms | Six months
  Respiratory symptoms

CONTACTS AND LOCATIONS:
Overall Officials: David CL Lam, MBBS,PhD,FCCP,FACP,FRCP(E), Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong Queen Mary Hospital, Hong Kong, Hong Kong